CLINICAL TRIAL: NCT00356148
Title: Phase IV Study of Determining the Efficacy of Ampicillin/Sulbactam Combination as Antibiotic Prophylaxis During Breast Cancer Surgery in Patients With a Body Mass Index (BMI) Over 25.
Brief Title: The Efficacy of Prophylactic Antibiotic Administration During Breast Cancer Surgery in Overweight Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Bahadir M. Gulluoglu, M.D., Prof Bahadir M Gulluoglu, MD, FACS, Marmara University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: MAR-YC-2003-0111
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast surgery; clean wound; overweight; prophylaxis; antibiotics
MeSH Terms: conditions — Breast Neoplasms; Overweight | interventions — sultamicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis Group (Active Comparator): patients who are BMI over 25 and receiving ampicillin/sulbactam prophylaxis
  Interventions: Drug: Ampicillin/Sulbactam
- No Prophylaxis Group (No Intervention): Patients who are BMI over 25 and do not receive antibiotic prophylaxis

INTERVENTIONS:
Drug: Ampicillin/Sulbactam — Ampicillin/Sulbactam 1 gr, once within onr hour before surgery
  Other Names: Ampisid 1 gr
  Arms: Prophylaxis Group

SUMMARY:
This is a single center trial to compare the rate of surgical site infection (SSI) in normal (BMI equal to or less than 25; Control Group)) and overweight (BMI over 25) women who are undergoing breast cancer surgery. The overweight patients are further randomized into two groups; in one group patients receive prophylactic antibiotics (ampicillin/sulbactam; Prophylaxis Group), in the other they do not (No Prophylaxis Group).

DETAILED DESCRIPTION:
CONTEXT Although breast surgery is regarded as clean surgery, the actual SSI rate is well above accepted range in various series. Retrospective studies showed BMI as one of the factors which may have caused increased SSI rate after breast cancer surgery. Yet, no prospective randomized study assessed the efficacy of chemoprophylaxis during breast surgery in overweight patients.

OBJECTIVE To compare the SSI rate between three groups of early stage breast cancer patients in which two are assigned according to randomization. First, patients are grouped into two according to their BMI. All patients (Control Group) with BMI equal to or below 25 do not receive any antibiotics as prophylaxis. Patients with a BMI above 25 are randomly assigned to receive a single dose prophylactic ampicillin /sulbactam combination before surgery (Prophylaxis Group) or not to receive chemoprophylaxis (No Prophylaxis Group).

DESIGN, SETTING AND PATIENTS Patient recruitment is still continuing after the study started in October 2003 in order to reach a sample size of 360 patients with BMI over 25. Advanced or distant metastatic stage, receiving neoadjuvant therapy, history of receiving antibiotics within prior 3 months, history of immunodeficiency, having a remote infection and history of reaction to treatment antibiotics are within the exclusion criteria.

INTERVENTIONS All patients are followed for 30 days postoperatively (once in a week at the original surgical unit). Patients and the investigator who inspects all wounds are blinded. Cost of SSI-related prophylaxis and treatments (including additional hospital visits after discharge, physician charges, additional antibiotics, wound management, other drugs and interventions etc) is calculated in each study group and compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Women at any age with early stage breast cancer (stage I-II) and American Society of Anesthesiologists (ASA) score of I-II.

Exclusion Criteria:

* Ductal carcinoma in situ (DCIS; stage 0 cancer),
* Advanced or distant metastatic stage,
* Receiving any neoadjuvant therapy,
* History of receiving any antibiotics within prior 3 months,
* History of immunodeficiency,
* Having a remote infection,
* History of reaction to study antibiotics,
* Denial of signing the consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2003-10; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir M Gulluoglu, MD, FACS, Study Chair — Marmara University School of Medicine, Department of General Surgery, Breast and Endocrine Surgery Unit
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Cunningham M, Bunn F, Handscomb K. Prophylactic antibiotics to prevent surgical site infection after breast cancer surgery. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005360. doi: 10.1002/14651858.CD005360.pub2. PMID 16625637
- [Derived] Gulluoglu BM, Guler SA, Ugurlu MU, Culha G. Efficacy of prophylactic antibiotic administration for breast cancer surgery in overweight or obese patients: a randomized controlled trial. Ann Surg. 2013 Jan;257(1):37-43. doi: 10.1097/SLA.0b013e31826d832d. PMID 23001082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a tertiary university teaching hospital between October 2003 and March 2010.
Pre-assignment Details: Patients having male gender, diagnosis of Stage 0, locally advanced or bilateral breast cancer, receiving neoadjuvant treatment, planning to undergo reconstructive surgery, having immunodeficiency, receiving antibiotics during previous one month, undergoing breast / axilla operation before randomization, denying to provide consent were excluded.
Period: Overall Study
Arm/Group | Prophylaxis Group | No Prophylaxis Group
Started | 189 | 183
Completed | 187 | 182
Not Completed | 2 | 1
Not completed — Reoperation within 30 days | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis Group | No Prophylaxis Group | Total
Number analyzed (Participants) | 189 | 183 | 372
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.1) | 56.9 (14.1) | 57.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 183 | 372
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Body Mass Index (BMI) Over 25 Who Developed Surgical Site Infection (SSI) in Groups Who Received Antibiotic Prophylaxis (Prophylaxis Group) and no Prophylaxis (No Prophylaxis Group).
Time Frame: 1 month
Population: Analysis was intent-to-treat
Measure: Number; unit: participants
Groups:
- No Prophylaxis Group: Patients who are BMI over 25 and not receive antibiotic prophylaxis
Arm/Group | Prophylaxis Group | No Prophylaxis Group
Number analyzed (Participants) | 187 | 182
participants | 9 | 25

2. Secondary Outcome: Overall SSI-related Prophylaxis and Treatment Cost in Patients With BMI Over 25 Who Received Prophylaxis (Prophylaxis Group) and Not (No Prophylaxis Group).
Time Frame: 1 month
Measure: Mean (Standard Error); unit: Monetary unit in Turkish Liras
Groups:
- No Prophylaxis Group: Patients who are BMI over 25 and not receiving antibiotic prophylaxis
Arm/Group | Prophylaxis Group | No Prophylaxis Group
Number analyzed (Participants) | 187 | 182
Monetary unit in Turkish Liras | 30 (5.6) | 13 (3.2)

ADVERSE EVENTS:
Arm/Group | Prophylaxis Group | No Prophylaxis Group
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/183
Other Adverse Events (participants affected / at risk) | 0/189 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No